CLINICAL TRIAL: NCT02392884
Title: A Cognitive Rehabilitation Program to Promote Treatment Adherence for Individuals Who Are HIV Positive With Mild Neurocognitive Difficulties
Brief Title: HIV Medication Adherence in Underserved Populations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Smith, Posstdoctoral Scientist, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00033072
Record Dates: First submitted 2015-03-10; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome
Keywords: Human Immunodeficiency Virus; Acquired Immunodeficiency Syndrome; Cognitive Rehabilitation; Minority Health; Vulnerable Populations; Underserved, Patients; Medication Adherence; Medication Compliance; Medication Non-compliance; Medication Persistence; Medication Non-Adherence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EON-MEM (Active Comparator): Intervention: Cognitive Rehabilitation and compensatory strategies will be taught to subjects to help them remember routes, viral load count, CD4 count, faces of providers and managing their schedules. Over the course of 5 visits, subjects will receive this intervention.
  Interventions: Behavioral: Cognitive Rehabilitation
- Compensatory Cognitive Training (Active Comparator): Cognitive Rehabilitation and physical reminders, such as calendars, smart phones, self-notes and other methods to help subjects remember to attend all medical appointments and take their HIV medication. Subject will be exposed to 5 sessions of this particular training.
  Interventions: Behavioral: Cognitive Rehabilitation
- Psychoeducation (No Intervention): The psychoeducation group, which aims to teach subjects the importance of taking medications and attending all doctor's appointment for HIV treatment. If you subjects are assigned to this group, they will be followed and receive the care generally followed for individuals with this condition.

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — Provide cognitive techniques and teach compensatory strategies that subjects can use to help them remember to attend appointments, take their medications regularly, increase attention (conversational and task) and concentration, increase cognitive flexibility, develop better problem-solving skills.
  Arms: Compensatory Cognitive Training; EON-MEM

SUMMARY:
The purpose of this study is to determine whether cognitive rehabilitation or psychoeducation impacts medication adherence in HIV-1 seropositive individuals.

DETAILED DESCRIPTION:
Although antiretroviral therapy (ART) has proven extremely effective in the treatment of HIV and AIDS, the ability to effectively combat the disease is inconsequential when individuals do not take their medication as prescribed and do not attend their scheduled medical appointments. Non-adherence to effective ART and medical visits is widespread in the United States, especially among ethnic minorities. A recent study indicated that patients who miss a medical appointment in the first year of an HIV diagnosis show over twice the mortality rate of patients who attended all visits. This study is developed to investigate the relationship between HIV Associated Neurocognitive Disorder (HAND) and adherence to HIV treatment among traditionally marginalized populations. Participants will be administered a brief neuropsychiatric screener. Participants will be randomly enrolled one of two cognitive rehabilitation programs so they may learn compensatory cognitive strategies to remain treatment adherent, or they will be receive psychoeducation concerning the importance of taking their medications and regularly attending medical appointments. Participants will be tracked and followed-up with regarding their treatment adherence in regular intervals over the course of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 and older.
* Able and willing to provide written informed consent.
* Diagnosed as HIV-seropositive by licensed enzyme-linked immunoabsorbent assay (ELISA) or HIV-seropositive by Western blot (WB).
* Diagnosed as HIV seropositive within the last two years.
* Willing and able to provide adequate information for locator purposes.

Exclusion Criteria:

* Under the age of 18.
* Have ever sustained a traumatic brain injury.
* Have an obvious psychological/psychiatric disorder that would invalidate the informed consent process, or otherwise contraindicate participation in the study.
* Have a learning disability where they cannot read or write pass the third grade level.
* Have an active substance dependence diagnosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Medication Adherence in 6 Months (adherence score) | 1,2, 3, 6 months
  Patients may experience an increase in treatment adherence. High scores indicate increased levels of adherence, while low scores reflect difficulties with treatment adherence.

SECONDARY OUTCOMES:
Change in Self Efficacy in 6 Months (subjective self-control score) | 1, 2, 3, 6 months
  Subjects may experience an increase in subjective self-control over their HIV treatment. High scores indicate high levels of perceived control over their treatment, while lower scores reflect a reduced amount of perceived self-efficacy over their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Smith, PsyD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Barclay TR, Hinkin CH, Castellon SA, Mason KI, Reinhard MJ, Marion SD, Levine AJ, Durvasula RS. Age-associated predictors of medication adherence in HIV-positive adults: health beliefs, self-efficacy, and neurocognitive status. Health Psychol. 2007 Jan;26(1):40-9. doi: 10.1037/0278-6133.26.1.40. PMID 17209696
- [Background] Berger BE, Ferrans CE, Lashley FR. Measuring stigma in people with HIV: psychometric assessment of the HIV stigma scale. Res Nurs Health. 2001 Dec;24(6):518-29. doi: 10.1002/nur.10011. PMID 11746080
- [Background] Chang L, Ernst T, Leonido-Yee M, Speck O. Perfusion MRI detects rCBF abnormalities in early stages of HIV-cognitive motor complex. Neurology. 2000 Jan 25;54(2):389-96. doi: 10.1212/wnl.54.2.389. PMID 10668700
- [Background] Chang L, Ernst T, Witt MD, Ames N, Gaiefsky M, Miller E. Relationships among brain metabolites, cognitive function, and viral loads in antiretroviral-naive HIV patients. Neuroimage. 2002 Nov;17(3):1638-48. doi: 10.1006/nimg.2002.1254. PMID 12414302
- [Background] Chesney MA. The elusive gold standard. Future perspectives for HIV adherence assessment and intervention. J Acquir Immune Defic Syndr. 2006 Dec 1;43 Suppl 1:S149-55. doi: 10.1097/01.qai.0000243112.91293.26. PMID 17133199
- [Background] Chesney MA, Ickovics JR, Chambers DB, Gifford AL, Neidig J, Zwickl B, Wu AW. Self-reported adherence to antiretroviral medications among participants in HIV clinical trials: the AACTG adherence instruments. Patient Care Committee & Adherence Working Group of the Outcomes Committee of the Adult AIDS Clinical Trials Group (AACTG). AIDS Care. 2000 Jun;12(3):255-66. doi: 10.1080/09540120050042891. PMID 10928201
- [Background] Contardo C, Black AC, Beauvais J, Dieckhaus K, Rosen MI. Relationship of prospective memory to neuropsychological function and antiretroviral adherence. Arch Clin Neuropsychol. 2009 Sep;24(6):547-54. doi: 10.1093/arclin/acp046. Epub 2009 Jul 31. PMID 19648150
- [Background] Crum NF, Riffenburgh RH, Wegner S, Agan BK, Tasker SA, Spooner KM, Armstrong AW, Fraser S, Wallace MR; Triservice AIDS Clinical Consortium. Comparisons of causes of death and mortality rates among HIV-infected persons: analysis of the pre-, early, and late HAART (highly active antiretroviral therapy) eras. J Acquir Immune Defic Syndr. 2006 Feb 1;41(2):194-200. doi: 10.1097/01.qai.0000179459.31562.16. PMID 16394852
- [Background] Fogarty L, Roter D, Larson S, Burke J, Gillespie J, Levy R. Patient adherence to HIV medication regimens: a review of published and abstract reports. Patient Educ Couns. 2002 Feb;46(2):93-108. doi: 10.1016/s0738-3991(01)00219-1. PMID 11867239
- [Background] Gonzalez JS, Hendriksen ES, Collins EM, Duran RE, Safren SA. Latinos and HIV/AIDS: examining factors related to disparity and identifying opportunities for psychosocial intervention research. AIDS Behav. 2009 Jun;13(3):582-602. doi: 10.1007/s10461-008-9402-4. Epub 2008 May 23. PMID 18498050
- [Background] Goujard C, Bernard N, Sohier N, Peyramond D, Lancon F, Chwalow J, Arnould B, Delfraissy JF. Impact of a patient education program on adherence to HIV medication: a randomized clinical trial. J Acquir Immune Defic Syndr. 2003 Oct 1;34(2):191-4. doi: 10.1097/00126334-200310010-00009. PMID 14526208
- [Background] Hinkin CH, Hardy DJ, Mason KI, Castellon SA, Lam MN, Stefaniak M, Zolnikov B. Verbal and spatial working memory performance among HIV-infected adults. J Int Neuropsychol Soc. 2002 May;8(4):532-8. doi: 10.1017/s1355617702814278. PMID 12030306
- [Background] Hinkin CH, Hardy DJ, Mason KI, Castellon SA, Durvasula RS, Lam MN, Stefaniak M. Medication adherence in HIV-infected adults: effect of patient age, cognitive status, and substance abuse. AIDS. 2004 Jan 1;18 Suppl 1(Suppl 1):S19-25. doi: 10.1097/00002030-200418001-00004. PMID 15075494
- [Background] Kumar V, Encinosa W. Effects of antidepressant treatment on antiretroviral regimen adherence among depressed HIV-infected patients. Psychiatr Q. 2009 Sep;80(3):131-41. doi: 10.1007/s11126-009-9100-z. Epub 2009 Apr 22. PMID 19387832
- [Background] Lovejoy TI, Suhr JA. The relationship between neuropsychological functioning and HAART adherence in HIV-positive adults: a systematic review. J Behav Med. 2009 Oct;32(5):389-405. doi: 10.1007/s10865-009-9212-9. Epub 2009 Mar 17. PMID 19291386
- [Background] Malta M, Magnanini MM, Strathdee SA, Bastos FI. Adherence to antiretroviral therapy among HIV-infected drug users: a meta-analysis. AIDS Behav. 2010 Aug;14(4):731-47. doi: 10.1007/s10461-008-9489-7. Epub 2008 Nov 20. PMID 19020970
- [Background] Mugavero MJ, Lin HY, Willig JH, Westfall AO, Ulett KB, Routman JS, Abroms S, Raper JL, Saag MS, Allison JJ. Missed visits and mortality among patients establishing initial outpatient HIV treatment. Clin Infect Dis. 2009 Jan 15;48(2):248-56. doi: 10.1086/595705. PMID 19072715
- [Background] Mugavero M, Ostermann J, Whetten K, Leserman J, Swartz M, Stangl D, Thielman N. Barriers to antiretroviral adherence: the importance of depression, abuse, and other traumatic events. AIDS Patient Care STDS. 2006 Jun;20(6):418-28. doi: 10.1089/apc.2006.20.418. PMID 16789855
- [Background] Nicastri E, Leone S, Angeletti C, Palmisano L, Sarmati L, Chiesi A, Geraci A, Vella S, Narciso P, Corpolongo A, Andreoni M. Sex issues in HIV-1-infected persons during highly active antiretroviral therapy: a systematic review. J Antimicrob Chemother. 2007 Oct;60(4):724-32. doi: 10.1093/jac/dkm302. Epub 2007 Aug 21. PMID 17715125
- [Background] Nieuwkerk PT, Oort FJ. Self-reported adherence to antiretroviral therapy for HIV-1 infection and virologic treatment response: a meta-analysis. J Acquir Immune Defic Syndr. 2005 Apr 1;38(4):445-8. doi: 10.1097/01.qai.0000147522.34369.12. PMID 15764962
- [Background] Oh DL, Sarafian F, Silvestre A, Brown T, Jacobson L, Badri S, Detels R. Evaluation of adherence and factors affecting adherence to combination antiretroviral therapy among White, Hispanic, and Black men in the MACS Cohort. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):290-3. doi: 10.1097/QAI.0b013e3181ab6d48. PMID 19521251
- [Background] Paasche-Orlow MK, Cheng DM, Palepu A, Meli S, Faber V, Samet JH. Health literacy, antiretroviral adherence, and HIV-RNA suppression: a longitudinal perspective. J Gen Intern Med. 2006 Aug;21(8):835-40. doi: 10.1111/j.1525-1497.2006.00527.x. PMID 16881943
- [Background] Power R, Koopman C, Volk J, Israelski DM, Stone L, Chesney MA, Spiegel D. Social support, substance use, and denial in relationship to antiretroviral treatment adherence among HIV-infected persons. AIDS Patient Care STDS. 2003 May;17(5):245-52. doi: 10.1089/108729103321655890. PMID 12816618
- [Background] Reynolds NR, Testa MA, Marc LG, Chesney MA, Neidig JL, Smith SR, Vella S, Robbins GK; Protocol Teams of ACTG 384, ACTG 731 and A5031s. Factors influencing medication adherence beliefs and self-efficacy in persons naive to antiretroviral therapy: a multicenter, cross-sectional study. AIDS Behav. 2004 Jun;8(2):141-50. doi: 10.1023/B:AIBE.0000030245.52406.bb. PMID 15187476
- [Background] Reynolds NR, Sun J, Nagaraja HN, Gifford AL, Wu AW, Chesney MA. Optimizing measurement of self-reported adherence with the ACTG Adherence Questionnaire: a cross-protocol analysis. J Acquir Immune Defic Syndr. 2007 Dec 1;46(4):402-9. doi: 10.1097/qai.0b013e318158a44f. PMID 18077832
- [Background] Safren SA, Otto MW, Worth JL, Salomon E, Johnson W, Mayer K, Boswell S. Two strategies to increase adherence to HIV antiretroviral medication: life-steps and medication monitoring. Behav Res Ther. 2001 Oct;39(10):1151-62. doi: 10.1016/s0005-7967(00)00091-7. PMID 11579986
- [Background] Santos CP, Felipe YX, Braga PE, Ramos D, Lima RO, Segurado AC. Self-perception of body changes in persons living with HIV/AIDS: prevalence and associated factors. AIDS. 2005 Oct;19 Suppl 4:S14-21. doi: 10.1097/01.aids.0000191485.92285.c7. PMID 16249648
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991;32(6):705-14. doi: 10.1016/0277-9536(91)90150-b. PMID 2035047
- [Background] Simoni JM, Kurth AE, Pearson CR, Pantalone DW, Merrill JO, Frick PA. Self-report measures of antiretroviral therapy adherence: A review with recommendations for HIV research and clinical management. AIDS Behav. 2006 May;10(3):227-45. doi: 10.1007/s10461-006-9078-6. PMID 16783535
- [Background] Turner BJ. Adherence to antiretroviral therapy by human immunodeficiency virus-infected patients. J Infect Dis. 2002 May 15;185 Suppl 2:S143-51. doi: 10.1086/340197. PMID 12001036
- [Background] van Servellen G, Carpio F, Lopez M, Garcia-Teague L, Herrera G, Monterrosa F, Gomez R, Lombardi E. Program to enhance health literacy and treatment adherence in low-income HIV-infected Latino men and women. AIDS Patient Care STDS. 2003 Nov;17(11):581-94. doi: 10.1089/108729103322555971. PMID 14746666
- [Background] Wagner GJ. Predictors of antiretroviral adherence as measured by self-report, electronic monitoring, and medication diaries. AIDS Patient Care STDS. 2002 Dec;16(12):599-608. doi: 10.1089/108729102761882134. PMID 12542933
- [Background] Woods SP, Moore DJ, Weber E, Grant I. Cognitive neuropsychology of HIV-associated neurocognitive disorders. Neuropsychol Rev. 2009 Jun;19(2):152-68. doi: 10.1007/s11065-009-9102-5. Epub 2009 May 22. PMID 19462243
- [Background] Reekie J, Mocroft A, Sambatakou H, Machala L, Chiesi A, van Lunzen J, Clumeck N, Kirk O, Gazzard B, Lundgren JD; EuroSIDA Study Group. Does less frequent routine monitoring of patients on a stable, fully suppressed cART regimen lead to an increased risk of treatment failure? AIDS. 2008 Nov 12;22(17):2381-90. doi: 10.1097/QAD.0b013e328317a6eb. PMID 18981778
- [Background] Lazo M, Gange SJ, Wilson TE, Anastos K, Ostrow DG, Witt MD, Jacobson LP. Patterns and predictors of changes in adherence to highly active antiretroviral therapy: longitudinal study of men and women. Clin Infect Dis. 2007 Nov 15;45(10):1377-85. doi: 10.1086/522762. Epub 2007 Oct 11. PMID 17968839
- [Background] Pellowski JA, Kalichman SC. Health behavior predictors of medication adherence among low health literacy people living with HIV/AIDS. J Health Psychol. 2016 Sep;21(9):1981-91. doi: 10.1177/1359105315569617. Epub 2015 Feb 20. PMID 25706334
- [Background] Pellowski JA, Kalichman SC, White D, Amaral CM, Hoyt G, Kalichman MO. Real-time medication adherence monitoring intervention: test of concept in people living with HIV infection. J Assoc Nurses AIDS Care. 2014 Nov-Dec;25(6):646-51. doi: 10.1016/j.jana.2014.06.002. Epub 2014 Jul 16. No abstract available. PMID 25043931
- [Background] Pellowski JA, Kalichman SC, Grebler T. Optimal Treatment Adherence Counseling Outcomes for People Living with HIV and Limited Health Literacy. Behav Med. 2016;42(1):39-47. doi: 10.1080/08964289.2014.963006. Epub 2014 Dec 13. PMID 25211524
- [Background] Kalichman S, Pellowski J, Chen Y. Requesting help to understand medical information among people living with HIV and poor health literacy. AIDS Patient Care STDS. 2013 Jun;27(6):326-32. doi: 10.1089/apc.2013.0056. Epub 2013 May 23. PMID 23701199
- [Background] Pellowski JA, Kalichman SC, Matthews KA, Adler N. A pandemic of the poor: social disadvantage and the U.S. HIV epidemic. Am Psychol. 2013 May-Jun;68(4):197-209. doi: 10.1037/a0032694. PMID 23688088
- [Background] Kalichman SC, Pellowski J, Kalichman MO, Cherry C, Detorio M, Caliendo AM, Schinazi RF. Food insufficiency and medication adherence among people living with HIV/AIDS in urban and peri-urban settings. Prev Sci. 2011 Sep;12(3):324-32. doi: 10.1007/s11121-011-0222-9. PMID 21607719
- [Background] Claborn KR, Meier E, Miller MB, Leffingwell TR. A systematic review of treatment fatigue among HIV-infected patients prescribed antiretroviral therapy. Psychol Health Med. 2015;20(3):255-65. doi: 10.1080/13548506.2014.945601. Epub 2014 Aug 11. PMID 25110152
- [Background] Marrazzo JM, del Rio C, Holtgrave DR, Cohen MS, Kalichman SC, Mayer KH, Montaner JS, Wheeler DP, Grant RM, Grinsztejn B, Kumarasamy N, Shoptaw S, Walensky RP, Dabis F, Sugarman J, Benson CA; International Antiviral Society-USA Panel. HIV prevention in clinical care settings: 2014 recommendations of the International Antiviral Society-USA Panel. JAMA. 2014 Jul 23-30;312(4):390-409. doi: 10.1001/jama.2014.7999. PMID 25038358
- [Background] Kalichman SC, Cherry C, Kalichman MO, Amaral C, White D, Grebler T, Eaton LA, Cruess D, Detorio MA, Caliendo AM, Schinazi RF. Randomized clinical trial of HIV treatment adherence counseling interventions for people living with HIV and limited health literacy. J Acquir Immune Defic Syndr. 2013 May 1;63(1):42-50. doi: 10.1097/QAI.0b013e318286ce49. PMID 23337369